CLINICAL TRIAL: NCT03876184
Title: Randomised Controlled Trial of the Alignment Efficiency and Coating Durability of Aesthetic Archwires
Brief Title: Alignment Efficiency and Coating Durability of Aesthetic Archwires
Acronym: RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Anis Kamaruddin, Principal investigator, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: USM/JEPeM/17010022
Record Dates: First submitted 2019-03-10; First posted 2019-03-15 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Tooth Movement
Keywords: tooth alignment; coating loss; color change; patient perception; aesthetic archwire
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The participants will select only one sealed envelope containing the archwires which has been labelled and coded without looking at other archwires. Both operators and participants are not informed of the brands of the coated archwires. The statistician will analyse the data based on the assigned codes. The codes will be broken by the principal investigator after the results have been produced.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- RMO FLi® Tooth-coloured superelastic Nickel Titanium (Experimental): This group has been allocated with upper and lower round 0.014" RMO FLi® Tooth-coloured superelastic Nickel Titanium aesthetic archwires for a duration of 8 weeks.
  Interventions: Other: Aesthetic archwires
- G&H G4 Tooth-coloured superelastic Nickel Titanium (Experimental): This group has been allocated with upper and lower round 0.014" G&H G4 Tooth-coloured superelastic Nickel Titanium aesthetic archwires for a duration of 8 weeks.
  Interventions: Other: Aesthetic archwires
- Orthocare Euroform® Cosmetic Tooth-coloured superelastic Nickel Titanium (Experimental): This group has been allocated with upper and lower round 0.014" Orthocare Euroform® Cosmetic Tooth-coloured superelastic Nickel Titanium aesthetic archwires for a duration of 8 weeks.
  Interventions: Other: Aesthetic archwires
- Conventional superelastic Nickel Titanium (Active Comparator): This group has been allocated with conventional upper and lower round 0.014" superelastic Nickel Titanium archwires for a duration of 8 weeks.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Aesthetic archwires — During bond-up, randomly allocated envelope will be opened and archwires will be ligated with elastomeric ligatures.After 4 weeks,the same archwires will be retied.Any fractured archwire will be recorded and discarded.The fractured wire will be replaced with conventional archwire and treatment continues.On the 2nd follow-up (at 8th week), the tested wires are collected, disinfected, dried and placed back in the allocated envelope.Upper and lower impressions will be taken.Questionnaires will be answered by participants.The trial ends and treatment continues as planned.Fractured archwire will be recorded and discarded.
  Arms: G&H G4 Tooth-coloured superelastic Nickel Titanium; Orthocare Euroform® Cosmetic Tooth-coloured superelastic Nickel Titanium; RMO FLi® Tooth-coloured superelastic Nickel Titanium
Other: Control group — During bond-up, randomly allocated envelope will be opened and archwires will be ligated with elastomeric ligatures.After 4 weeks,the same archwires will be retied.Any fractured archwire will be recorded and discarded.The fractured wire will be replaced with conventional archwire and treatment continues.On the 2nd follow-up (at 8th week), the tested wires are collected, disinfected, dried and placed back in the allocated envelope.Upper and lower impressions will be taken.This group will not answer the questionnaire.The trial ends and treatment continues as planned.Fractured archwire will be recorded and discarded.
  Arms: Conventional superelastic Nickel Titanium

SUMMARY:
This study investigates the efficiency of orthodontic aesthetic archwires which are coated with tooth-colored materials and the durability of the coatings after being used. Theoretically, the coatings provide excellent aesthetics throughout treatment and faster tooth alignment. However, from our clinical experience, these claims are the opposite. Cracks and ruptures as well as archwire fractures have been noted. Therefore, it is presumed that the aesthetic archwires may not be any different from the conventional uncoated archwires.

DETAILED DESCRIPTION:
The development of superelastics nickel titanium (SE NiTi) has overcome problems with previous aligning archwires. This archwire is deemed to be the gold standard aligning archwire for Straight Wire® system due to its shape memory effect, high elasticity and low permanent deformation which delivers continuous force for orthodontic tooth alignment. The only drawbacks of this wire type are it is expensive, have high frictional resistance (Kapila et al., 1990) and is associated with hypersensitivity reaction in nickel allergic patients (Bass et al., 1993).

Development of teflon or polytetrafluoroethylene (PTFE) which is anti-adherent and possesses aesthetic property had been used as orthodontic bracket, archwire and ligature coating. This polymer consists of synthetic fluorine-containing resin or epoxy resin composed mainly of polytetrafluoroethylyene to simulate tooth colour. The polymeric chain with good mechanical stability had been shown to reduce the frictional resistance between bracket-archwire interface and when used as archwire ligature (Farronato et al., 2012, De Franco et al., 1995). PTFE-coated brackets were reported to minimise the formation of biofilm during treatment which can reduce the risk of enamel decalcification (Demling et al., 2010). Furthermore, the coated aesthetic archwires have potential to obviate any allergic reaction during orthodontic treatment in patients with known hypersensitivity to nickel alloy.

Manufacturers have claimed that the aesthetic archwires available in the market have good color stability (remains unchanged for 6 to 8-week duration), good coating durability and low friction, allowing faster tooth movement. However, to our experience, these claims are the opposite.

As these aesthetic archwires are much more expensive than the conventional superelastic nickel titanium, it is therefore important to establish a clinical data to allow clinicians and patients to make a justifiable choice on treatment and develop further research in this area.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 11 years old and above in permanent dentition with all teeth from upper and lower 6 - 6 are present, tooth apices are closed
* Patients who require complete bond-up with upper and lower pre-adjusted edgewise bracket system, MBT prescription with bracket slot size 0.022"
* Able to give consent* *Assent form is required for children below 18 years of age

Exclusion Criteria:

* Patients with cleft lip and palate and other craniofacial deformities and syndromes
* Patients with medical problems / medications that can influence rate of tooth movement
* Teeth blocked out of the arch / ectopic teeth not allowing bracket placement and ligation at bond-up
* Hypodontia with more than one tooth missing in any quadrant
* Have had orthodontic treatment before

Min Age: 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-01-31 (Actual)

PRIMARY OUTCOMES:
Alignment efficiency | 8 weeks
  The tooth irregularity between pre- and post-experiment dental casts are measured in millimetres. The difference between the two measurement will be calculated in percentage.

SECONDARY OUTCOMES:
Coating loss | 8 weeks
  The amount of coating loss between the used and unused archwires will be measured in percentage.
Color change | 8 weeks
  The difference in colour (colour change) between used and unused archwires will be measured in CIE L* a* b* colour space units.
Participant perception towards aesthetic archwires | 8 weeks
  Patient perception will be assessed using oral aesthetic subjective impact scale (OASIS) questionnaires after the use of aesthetic archwires (at week 8). The cumulative score will be used to determine the perception (14 and below = positive perception; 15 and above = negative perception).

CONTACTS AND LOCATIONS:
Overall Officials: Anis F Kamaruddin, MOrth, Principal Investigator — Advanced Medical & Dental Institute
Locations (3):
- Malaysia (3):
  - School of Dental Sciences, Kubang Kerian, Kelantan
  - Advanced Medical & Dental Institute, Kepala Batas, Pulau Pinang
  - Desa Murni Dental Clinic, Permatang Pauh, Pulau Pinang

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in publication
Supporting Information: SAP, ICF
Time Frame: 6 months after publication.
Access Criteria: Describe by what Access criteria IPD and any additional supporting information will be shared through email with other researchers. Principal investigator will review requests prior to data sharing.

REFERENCES:
- [Background] Bass JK, Fine H, Cisneros GJ. Nickel hypersensitivity in the orthodontic patient. Am J Orthod Dentofacial Orthop. 1993 Mar;103(3):280-5. doi: 10.1016/0889-5406(93)70009-D. PMID 8456786
- [Background] Kapila S, Angolkar PV, Duncanson MG Jr, Nanda RS. Evaluation of friction between edgewise stainless steel brackets and orthodontic wires of four alloys. Am J Orthod Dentofacial Orthop. 1990 Aug;98(2):117-26. doi: 10.1016/0889-5406(90)70005-W. PMID 2378317
- [Background] Farronato G, Maijer R, Caria MP, Esposito L, Alberzoni D, Cacciatore G. The effect of Teflon coating on the resistance to sliding of orthodontic archwires. Eur J Orthod. 2012 Aug;34(4):410-7. doi: 10.1093/ejo/cjr011. Epub 2011 Apr 8. PMID 21478301
- [Background] Demling A, Elter C, Heidenblut T, Bach FW, Hahn A, Schwestka-Polly R, Stiesch M, Heuer W. Reduction of biofilm on orthodontic brackets with the use of a polytetrafluoroethylene coating. Eur J Orthod. 2010 Aug;32(4):414-8. doi: 10.1093/ejo/cjp142. Epub 2010 Feb 5. PMID 20139131
- [Background] De Franco DJ, Spiller RE Jr, von Fraunhofer JA. Frictional resistances using Teflon-coated ligatures with various bracket-archwire combinations. Angle Orthod. 1995;65(1):63-72; discussion 73-4. doi: 10.1043/0003-3219(1995)0652.0.CO;2. PMID 7726464